CLINICAL TRIAL: NCT03119207
Title: Creating Naptime: An Overnight, Non-Pharmacologic Intensive Care Unit Sleep Promotion Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1112009428; P20NR014126 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Sleep
Keywords: ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Naptime Participants (Experimental): The participants will undergo the Naptime Protocol. The study team will provide a 4 hour period nightly during which patient room activity, light levels and noise levels will be decreased. The team will monitor the changes in the number and quality of these disruptions and to monitor the changes in patient sleep and outcome following our intervention.
  Interventions: Behavioral: Naptime Protocol
- Control Participants (No Intervention): Naptime will not be enforced. Patient room activity, light levels and noise levels are monitored. Standard care will be provided. During the intervention period patients are randomized to either control or naptime.
- Baseline Participants (No Intervention): Prior to the intervention period, baseline patients under usual care are monitored. Naptime will not be enforced. Patient room activity, light levels and noise levels are monitored.

INTERVENTIONS:
Behavioral: Naptime Protocol — Between midnight and 4:00 every attempt will be made to limit staff entrance into the patient room.
  Arms: Naptime Participants

SUMMARY:
Specific Aims:

1. Quantify baseline patient room disruptions in the medical ICU during the proposed nocturnal Naptime .

   1. Obtain baseline light and noise levels in selected medical ICU study rooms.
   2. Obtain baseline activity level levels in selected medical ICU study rooms.
   3. Assess baseline information regarding nursing experience, prior training / beliefs regarding sleep promotion in the medical ICU
2. Assess the feasibility of instituting a 4 hour (Midnight to 4:00 AM) nocturnal Naptime with minimization of patient interaction via tracking of differences in patient room activity, light and noise levels in control versus intervention patients.

   Secondary Aim
3. Examine the associations between Naptime provision and patient sleep quality.

DETAILED DESCRIPTION:
The effects of poor sleep are dauntingly pleiotropic. Inasmuch as sleep deprivation can behaviorally and physiologically mimic delirium in the ICU, there is concern that sleep deprived ICU patients are at risk for the increased mortality, longer hospital stays and worsened physical and mental outcomes of hospitalized patients who experience delirium during their admission. Furthermore, lack of sleep has been associated with decrements in FEV1, FVC and maximal inspiratory pressure in non-ICU COPD patients, increases in respiratory muscle fatigue in healthy volunteers and blunted response to hypercapnea in healthy volunteers. Finally, theoretical concerns exist regarding sleep loss putting patients at risk for prolonged bedrest, adverse cardiovascular events, derangement of metabolism and endocrine function as well as immune suppression; though supported by animal models and brief studies in healthy volunteers, no ICU data exists.

ELIGIBILITY:
Inclusion Criteria:

* All MICU admissions age 18 and older who are admitted no less than 6 hours and no more than 48 hours prior to intended start of the next potential Naptime (midnight start).

Exclusion Criteria:

* Patients who are "boarding" from other intensive care units at Yale New Haven Hospital; these patients are not cared for by our providers and would not be subject to our protocols.
* Patients without an identifiable surrogate who cannot consent for themselves.
* Comfort care only patients
* Patients undergoing the hypothermia protocol.
* Patients enrolled in the MIND*USA delirium study.
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-11-04 (Actual); Primary Completion 2014-06-22 (Actual); Study Completion 2014-06-22 (Actual)

PRIMARY OUTCOMES:
Sound Level | Day 1-3 following study enrollment
  Sound levels in the patient room will be monitored overnight for the three nights following enrollment. Sound level recordings will include 8:00 PM to 12:00PM (noon) on the following day to track the Naptime period (12:00 AM/midnight to 4:00 AM) and adjacent control periods.
Light Level | Day 1-3 following study enrollment
  Light levels in the patient room will be monitored overnight for the three nights following enrollment. Light level recordings will include 8:00 PM to 12:00PM (noon) on the following day to track the Naptime period (12:00 AM/midnight to 4:00 AM) and adjacent control periods.
Number of Room Entrances | Day 1-3 following study enrollment
  The number of room entrances will be monitored overnight for the three nights following enrollment via videography of the room door. Videography will include 8:00 PM to 12:00PM (noon) on the following day to track the Naptime period (12:00 AM/midnight to 4:00 AM) and adjacent control periods.
Length of Room Entrances | Day 1-3 following study enrollment
  The length of room entrances will be monitored overnight for the three nights following enrollment via videography of the room door. Videography will include 8:00 PM to 12:00PM (noon) on the following day to track the Naptime period (12:00 AM/midnight to 4:00 AM) and adjacent control periods.
Length of Rest Periods between Room Entrances | Day 1-3 following study enrollment
  The length of rest periods between room entrances will be monitored overnight for the three nights following enrollment via videography of the room door. Videography will include 8:00 PM to 12:00PM (noon) on the following day to track the Naptime period (12:00 AM/midnight to 4:00 AM) and adjacent control periods.

SECONDARY OUTCOMES:
RCSQ score | Day 1-3 following study enrollment
  The Richards Campbell Sleep Questionnaire will be administered to all patients and their primary overnight nurses to evaluate sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Knauert, MD, PhD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No